CLINICAL TRIAL: NCT04104841
Title: School-Based Depression Prevention for Adolescents With ADHD
Acronym: BEAMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MH117086; R34MH117086 (NIH)
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Attention Deficit Hyperactivity Disorder; Depressive Symptoms
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Depression | interventions — Schools

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behaviorally Enhancing Adolescents' Mood in Schools (BEAMS) (Experimental): 8-session modified behavioral activation program
  Interventions: Behavioral: Behaviorally Enhancing Adolescents' Mood in Schools
- Usual Care (Active Comparator): Referrals to usual care
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Behaviorally Enhancing Adolescents' Mood in Schools — 8-session modified behavioral activation intervention
  Arms: Behaviorally Enhancing Adolescents' Mood in Schools (BEAMS)
Behavioral: Usual Care — Referral to school mental health provider, social worker, or community care.
  Arms: Usual Care

SUMMARY:
The purpose of this study is to develop a modified behavioral activation program in adolescents with ADHD to be implemented by school mental health providers in an urban, low-income school district. Subsequently the investigators will examine its effectiveness in reducing depressive symptoms and improving emotion regulation and reward responsivity, compared to usual care.

DETAILED DESCRIPTION:
Children with ADHD are at elevated risk for depression in adolescence and young adulthood, and this comorbidity is associated with far greater impairment than either disorder alone, including higher rates of inpatient hospitalization and increased risk for suicidal ideation and behavior. Despite these adverse outcomes, existing evidence-based interventions for ADHD have not demonstrated effects in reducing depressive symptoms nor do established depression prevention programs work as well for adolescents with ADHD. Reward responsivity (RR) and emotion regulation (ER) are two key factors demonstrated to mediate the association between ADHD and depression and are thus key targets for prevention. In an effort to address the gap between access and utilization of mental health care, which is especially stark among adolescents with ADHD, the investigators aim to develop and test a modified behavioral activation prevention program [Behaviorally Enhancing Adolescents' Mood in Schools (BEAM-S)] that incorporates modules to directly target these purported mechanisms. In line with the Deployment-Focused Model of Intervention Development and Testing, the investigators will develop a program that can be easily implemented and sustainable in the high school setting as delivered by school mental health staff that reduces depression and improves overall functioning in adolescents with ADHD, by way of improving RR and ER. As a first step, the investigators will conduct focus groups with community stakeholders (e.g., school mental health providers, school administration, adolescents, parents, teachers) to develop an acceptable and sustainable selected and indicated prevention program for school staff to utilize. The investigators will then initially train school staff to deliver this prevention program via to pilot the intervention for implementation of the prevention program in a case series to evaluate preliminary feasibility. The investigators will then conduct a stage 1 RCT with a hybrid-type 1 implementation effectiveness design in three high schools where adolescents will be randomized to either the BEAM-S condition (n= 54) or treatment as usual (n = 54). Finally, qualitative and quantitative data from aims 1-3 will be used to prepare final procedures for a future large-scale effectiveness trial R01 (aim 4).

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in a participating Baltimore City Public High School
* DSM-5 Diagnosis of attention-deficit/hyperactivity disorder (ADHD)
* Depressive symptoms above T=65 on the Children's Depression Inventory (CDI)

Exclusion Criteria:

* History of seizures or neurological problems
* DSM-diagnosis of Pervasive Developmental Disorder
* Full scale IQ below 70
* Current depressive symptoms or active suicidality at severe levels where more intensive services would be warranted

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-07-11 (Actual)

PRIMARY OUTCOMES:
Children's Depression Inventory, 2nd Edition (CDI-2) | After the 8-week preventive intervention
  Adolescent and parent reported depressive symptoms
Children's Depression Inventory, 2nd Edition (CDI-2) | 4-week follow-up
  Adolescent and parent reported depressive symptoms
Children's Depression Inventory, 2nd Edition (CDI-2) | 12-week follow-up
  Adolescent and parent reported depressive symptoms

SECONDARY OUTCOMES:
Affective Reactivity Index | After the 8-week preventive intervention
  Adolescent and parent reported irritability
Affective Reactivity Index | 4-week follow-up
  Adolescent and parent reported irritability
Affective Reactivity Index | 12-week follow-up
  Adolescent and parent reported irritability
Suicide Behavior Questionnaire | After the 8-week preventive intervention
  Adolescent reported suicidal thoughts and behaviors
Suicide Behavior Questionnaire | 4-week follow-up
  Adolescent reported suicidal thoughts and behaviors
Suicide Behavior Questionnaire | 12-week follow-up
  Adolescent reported suicidal thoughts and behaviors
Emotion Regulation Checklist | After the 8-week preventive intervention
  Parent reported emotion dysregulation
Emotion Regulation Checklist | 4-week follow-up
  Parent reported emotion dysregulation
Emotion Regulation Checklist | 12-week follow-up
  Parent reported emotion dysregulation
Difficulties in Emotion Regulation | After the 8-week preventive intervention
  Adolescent reported emotion dysregulation
Difficulties in Emotion Regulation | 4-week follow-up
  Adolescent reported emotion dysregulation
Difficulties in Emotion Regulation | 12-week follow-up
  Adolescent reported emotion dysregulation
Mirror Tracing Persistence Task | After the 8-week preventive intervention
  Emotion regulation behavioral task
Mirror Tracing Persistence Task | 4-week follow-up
  Emotion regulation behavioral task
Mirror Tracing Persistence Task | 12-week follow-up
  Emotion regulation behavioral task
Tripartite Pleasure Inventory | After the 8-week preventive intervention
  Adolescent reported reward responsiveness
Tripartite Pleasure Inventory | 4-week follow-up
  Adolescent reported reward responsiveness
Tripartite Pleasure Inventory | 12-week follow-up
  Adolescent reported reward responsiveness
Reward Probability Index | After the 8-week preventive intervention
  Measure of adolescent reported environmental reward
Reward Probability Index | 4-week follow-up
  Measure of adolescent reported environmental reward
Reward Probability Index | 12-week follow-up
  Measure of adolescent reported environmental reward
Behavioral Activation for Depression Scale | After the 8-week preventive intervention
  Adolescent reported measure of behavioral activation and avoidance
Behavioral Activation for Depression Scale | 4-week follow-up
  Adolescent reported measure of behavioral activation and avoidance
Behavioral Activation for Depression Scale | 12-week follow-up
  Adolescent reported measure of behavioral activation and avoidance
Balloon Analog Risk Task | After the 8-week preventive intervention
  Positive reinforcement
Balloon Analog Risk Task | 4-week follow-up
  Positive reinforcement
Balloon Analog Risk Task | 12-week follow-up
  Positive reinforcement
Impairment Rating Scale | After the 8-week preventive intervention
  Parent- and teacher- report of global impairment
Impairment Rating Scale | 4-week follow-up
  Parent- and teacher- report of global impairment
Impairment Rating Scale | 12-week follow-up
  Parent- and teacher- report of global impairment

CONTACTS AND LOCATIONS:
Overall Officials: Michael Meinzer, PhD, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland, College Park, Maryland, United States